CLINICAL TRIAL: NCT03752645
Title: Effect of Red Light Rhinophototherapy on Nasal Patency in Patients With Allergic Rhinitis
Brief Title: Subjects With Clinical Diagnosis of Allergic Rhinitis Were Randomly Divided Into 2 Groups, With Patients in One Group Given One Treatment Session of Red Light Rhinophototherapy, Followed by Medical Treatment. Those in the Second Group Were Treated With Medical Treatment Only.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CF18014A#1
Record Dates: First submitted 2018-11-17; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Allergic Rhinitis; Phototherapy
Keywords: acoustic rhinometry; active anterior rhinomanometry; allergic rhinitis; red light rhinophototherapy
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Transverse Many Channels Laser Instrument
  Interventions: Device: Transverse Many Channels Laser Instrument
- control (No Intervention)

INTERVENTIONS:
Device: Transverse Many Channels Laser Instrument — The device consists of a control box and 4 sets of two light-emitting nasal probes. Prior to treatment, each patient put on a pair of black tinted glasses, and had the nasal probes gently placed into both nostrils. A turn-on switch on the control box activated the probe and the timer was set at 15 minutes during which time 36 J of light energy was delivered to each nostril.
  Arms: intervention

SUMMARY:
To investigate the short-term effects of red light rhinophototherapy on nasal patency in patients with a clinical diagnosis of allergic rhinitis using both active anterior rhinomanometry and acoustic rhinometry.

DETAILED DESCRIPTION:
Patients experiencing moderate to severe symptoms of allergic rhinitis (AR)were collected. The clinical diagnosis of AR was established when patients presented themselves with a history and physical examination consistent with an allergic cause. Each candidate possessed at least one of the following symptoms: nasal congestion, runny nose, itchy nose, or sneezing. All patients underwent a specific IgE test against the common perennial inhaled allergens found in Taiwan (house dust mites, molds, cats, dogs and cockroaches) to confirm the diagnosis of AR. However, these results did not exclude the patients from this study because only a few allergens were tested. The severity of the rhinitis symptoms was assessed through use of a standardized score scale (1). A score of 0 (no symptoms), 1 (mild symptoms), 2 (moderate symptoms), to 3 (severe symptoms) was used to evaluate the severity of nasal congestion, runny nose, itchy nose, and sneezing. Patients receiving a total score of 4 or more were enrolled in the study. Patients with age below 20 years old, severe nasal septum, rhinosinusitis and nasal polyposis were excluded from the study. Those who had a history of immunodeficiency or previous sinus surgery, suffered from an upper respiratory tract infection, or took oral corticosteroids within a month prior to the study were also excluded.

Eligible patients were randomly divided into 2 groups. Randomization assignments were generated by an independent statistician. Patients in the study group were treated with one treatment session of red light rhinophototherapy (RLRPT) (40mW/nostril for 15 minutes) at the outpatient clinic after completing a nasal patency test using both active anterior rhinomanometry and acoustic rhinometry. Upon completing RLRPT treatment, patients took a rest for 30 minutes. They were then asked about the severity of their rhinitis symptoms, and as to whether the overall level of change in those rhinitis symptoms was worse, unchanged, slightly improved, much improved or cured. Patients were also questioned about any adverse events of RLRPT before undergoing another nasal patency test. Finally, medical treatment involving an intranasal steroid (mometasone furoate nasal spray, 4 sprays, once a day), along with an oral antihistamine (levocetirizine 5 mg qd) was given for continued management of AR. Questions regarding the severity of each patient's rhinitis symptoms, the overall change in their rhinitis symptoms and any adverse events from RLRPT were asked via telephone communication 2 days later. Patients in the active control group were medically treated with an intranasal steroid (mometasone furoate nasal spray, 4 sprays, once a day), along with an oral antihistamine (levocetirizine 5 mg qd). Telephone calls were placed 2 days later in order to evaluate the severity of each patient's rhinitis symptoms, along with any overall change in rhinitis symptoms.

The device used for RLRPT was the Transverse Many Channels Laser Instrument (Transverse, Ind, Co., Ltd., Taipei, Taiwan). It uses a red gallium-aluminum-arsenide laser with wavelengths of 660+10 nm as a light source. The laser has a maximum power of 40 mW. The device consists of a control box and 4 sets of two light-emitting nasal probes. Prior to treatment, each patient put on a pair of black tinted glasses, and had the nasal probes gently placed into both nostrils. A turn-on switch on the control box activated the probe and the timer was set at 15 minutes during which time 36 J of light energy was delivered to each nostril.

The nasal patency was objectively measured by both active anterior rhinomanometry and acoustic rhinometry. Anterior active rhinomanometry was performed according to the guidelines of the International Committee on Standardization of Rhinomanometry using a NR6 Rhinomanometer (GM Instruments, Ltd., Kilwinning, UK). All patients remained seated for 30 minutes to adapt to the hospital environment prior to testing. A face mask was worn tightly. The examination was performed during quiet breathing with a closed mouth, while the patient was in an upright sitting position. For each nostril, inspiratory nasal resistance was calculated over four inspiratory-expiratory cycles at a fixed pressure of 150 Pascal. Both the total nasal airflow resistance in Pa/cm3/s, and nasal airflow in cm3/s (sum of left and right) during inspiration were recorded.

An A1 Acoustic Rhinometer (GM Instruments, Ltd., Kilwinning, UK) was used to measure the geometry of the nasal cavity. All patients remained seated for at least 20 minutes in order to acclimatize to the hospital environment before testing. The nose piece was positioned parallel to the sagittal plane of the head at a 45° angle to the coronal plane, and was applied to produce an acoustic seal without distorting the outer nose. Patients were asked to hold their breath and avoid swallowing during the acquisition of the acoustic data. Three consecutive readings were taken to calculate an average value. An entire average acoustic rhinometry curve was generated for each nasal cavity. Acoustic data included: 1) the first minimal cross-sectional area (MCA1, cm2), 2) the second minimal cross sectional area (MCA2, cm2), 3) the volume between the tip of the nosepiece and 3.0 cm into the nasal cavity (V03, cm3), and 4) the volume of the nasal cavity between 2.0 and 5.0 cm from the tip of the nosepiece (V25, cm3). We used the average value of both sides to represent the data.

ELIGIBILITY:
Inclusion Criteria:

* Patients experiencing moderate to severe symptoms of allergic rhinitis
* Patients possessing at least one of the following symptoms: nasal congestion, runny nose, itchy nose, or sneezing
* Patients whose physical examination showing clear rhinorrhea, nasal congestion, pale discoloration of the nasal mucosa, or red and watery eyes

Exclusion Criteria:

* Patients with age below 20 years old
* Patients with severe nasal septum, rhinosinusitis and nasal polyposis
* Patients who had a history of immunodeficiency or previous sinus surgery
* Patients who suffered from an upper respiratory tract infection
* Patients who took oral corticosteroids within a month prior to the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in nasal resistance and nasal flow after red light Change from baseline in nasal resistance and nasal flow after red light rhinophototherapy | before and 30 minutes after red light rhinophototherapy
  To compare the change from baseline in nasal resistance and nasal flow 30 minutes after red light rhinophototherapy by using active anterior rhinomanometry
Change from baseline in the first and second minimal cross sectional area, and the volumes between the tip and 3.0 cm from the tip of the nosepiece and between 2.0 and 5.0 cm from the tip of the nosepiece after red light rhinophototherapy | before and 30 minutes after red light rhinophototherapy
  To compare the change from baseline in the first minimal cross sectional area of the nasal cavity, the second minimal cross sectional area of the nasal cavity, the nasal volume between the tip of the nosepiece and 3.0 cm into the nasal cavity, and the nasal volume of the nasal cavity between 2.0 and 5.0 cm from the tip of the nosepiece 30 minutes after red light rhinophototherapy by using acoustic rhinometry

SECONDARY OUTCOMES:
rhinitis symptoms | before red light rhinophototherapy, and 30 minutes and 2 days after red light rhinophototherapy
  The severity of the rhinitis symptoms was assessed through use of a standardized score scale (1). A score of 0 (no symptoms), 1 (mild symptoms), 2 (moderate symptoms), to 3 (severe symptoms) was used to evaluate the severity of nasal congestion, runny nose, itchy nose, and sneezing.

CONTACTS AND LOCATIONS:
Overall Officials: Rong-San Jiang, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Jiang RS, Wang JJ. Effect of Red Light Rhinophototherapy on Nasal Patency in Patients with Allergic Rhinitis. Int J Otolaryngol. 2018 Dec 17;2018:6270614. doi: 10.1155/2018/6270614. eCollection 2018. PMID 30647740